CLINICAL TRIAL: NCT05582720
Title: Development of Innovative Functional Meat Analogues Using Alternative Sources of Plant Proteins and Novel Technologies
Brief Title: Cardioprotective Properties of Vegan Burger
Acronym: VeganBurger
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harokopio University (Other)
Collaborators: Hellenic Catering S.A. (Unknown); Laboratory of Design and Process Analysis, School of Chemical Engineering, National Technical University of Athens (Unknown); Laboratory of Biotechnology, Department of Biological Applications & Technology, University of Ioannina (Unknown); European Regional Development Fund (Other)
Responsible Party: Principal Investigator, Tzortzis Nomikos, Associate Professor of Biochemistry, Harokopio University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Γ-3047/17-06-2021
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Cardiometabolic Health
Keywords: read meat; meat analogues; burger; vegan burger; dietary intervention; plant proteins; inflammation; oxidative stress; thrombosis; cardioprotection
MeSH Terms: conditions — Inflammation; Thrombosis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional burger group (Active Comparator): This arm will consume 2 portions (each 120 g cooked) of conventional burger per week for a 4-week period.
  Interventions: Behavioral: Conventional burger
- Vegan burger group (Experimental): This arm will consume 2 portions (each 120 g cooked) of vegan burger per week for a 4-week period.
  Interventions: Behavioral: Vegan burger

INTERVENTIONS:
Behavioral: Conventional burger — Participants initially randomized to this intervention arm will be provided with a total of 8 conventional burgers and will be asked to consume them twice weekly for 4 weeks. Conventional burgers will be produced by Hellenic Catering S.A. using standard procedures. Participants will also be instructed to maintain their usual dietary intake, physical activity level, prescribed medications and dietary supplements, as well as to refrain from any weight loss effort during the intervention. After a 2-week wash-out period (no burger consumption), participants will cross over to the other intervention arm.
  Arms: Conventional burger group
Behavioral: Vegan burger — Participants initially randomized to this intervention arm will be provided with a total of 8 vegan burgers and will be asked to consume them twice weekly for 4 weeks. Vegan burgers will be produced by Hellenic Catering S.A. using novel technologies. Participants will also be instructed to maintain their usual dietary intake, physical activity level, prescribed medications and dietary supplements, as well as to refrain from any weight loss effort during the intervention. After a 2-week wash-out period (no burger consumption), participants will cross over to the other intervention arm.
  Arms: Vegan burger group

SUMMARY:
Several studies over the last decades have demonstrated the important role of nutrition in the development of chronic diseases, such as cardiovascular disease and cancer. One dietary component that has been in the center of scientific research is red meat and processed meat (e.g., cold cuts, sausages, burgers). Burger, in particular, is one of the most popular red meat products and its consumption has increased rapidly in recent years due to the expansion of fast-food restaurants, its wide availability and its low price. However, due to its high animal fat content which is mostly saturated and high degree of processing, its nutritional value and the safety of its long-term high consumption have been questioned. The wide acceptance of burger by the general population, combined with the perception that it is a "burdensome" food for health, makes it an ideal subject for interventions aiming at modifying its nutritional value without downgrading its organoleptic characteristics and increasing its cost. Such an approach could be applied to the meat industry in order to develop innovative, functional meat analogues of high nutritional and organoleptic value, which could find acceptance by both meat-eating and vegetarian/vegan populations. Therefore, the aim of the present double-blind, randomized, crossover clinical trial is to explore the potential cardioprotective properties of "vegan burger", a novel meat analogue developed through the substitution of animal proteins and lipids with plant-based constituents using innovative technologies, against the conventional animal-based burger, in apparently healthy volunteers.

DETAILED DESCRIPTION:
The nutritional value and health effects of red meat and processed meat products (e.g., cold cuts, sausages, burgers) remain the object of intense research and scientific controversy in the fields of Nutrition and Food Science. Red meat is a rich source of macronutrients (e.g., proteins of high biological value) and several micronutrients (e.g., iron), and a food group particularly appealing to consumers. However, in recent years there has been an increase in the total consumption of red meat and processed meat products in developed countries, which has been associated with both increased risk of chronic diseases (e.g., cardiovascular diseases, obesity, diabetes mellitus, various types of cancer and autoimmune diseases) and increased total mortality. The aggravating effect of red meat consumption on health is likely attributed to its increased content of saturated fatty acids, which have been associated with the occurrence of insulin resistance, dyslipidemia, and disturbances in the intestinal microbiota, as well as other components produced during its processing (e.g., oxidized forms of fat, heterocyclic amines, polycyclic aromatic hydrocarbons), which can trigger mechanisms of inflammation, oxidative stress and carcinogenesis, and further contribute to the pathogenesis of cardiometabolic and neoplastic diseases. Based on the available research data, scientific associations and health organizations at the local and international level recommend limiting the consumption of red meat and meat products and replacing them with products of plant origin in the context of adopting a balanced health-promoting diet and reducing the risk of chronic cardiometabolic disorders in the general population.

Burger is one of the most popular meat products and its consumption has increased rapidly in recent years due to the expansion of fast-food restaurants, its wide availability and its low price. However, due to its high content in animal fat, which is mostly saturated, its nutritional value and the safety of its long-term high consumption have been questioned. The wide acceptance of burger by the general population, combined with the perception that it is a "burdensome" food for health, makes it an ideal subject for interventions aiming at modifying its nutritional value without simultaneously degrading its organoleptic characteristics and increasing its cost. Such an approach could be applied to the meat industry in order to develop innovative, functional meat analogues of high nutritional value, which could also find acceptance by meat-eating populations. The challenges in this direction are many, such as the reduction of lipids and/or the replacement of saturated fatty acids with other health-beneficial lipids without degrading the texture and taste of the product, and the replacement of animal proteins with plant proteins. Until now, the majority of commercially available meat analogs are made from soy protein or gluten. However, protein products have also been developed from other raw materials, including vegetables and legumes (e.g., peas and chickpeas). In addition, protein products from fungi and bacteria are available, which are suitable for reproducing the taste and texture of meat. Regarding fat, various ingredients have also been explored as substitutes for animal fat, such as dietary fiber and vegetable oils.

The aim of the present study is to explore the potential cardio-protective effects of an innovative burger of high nutritional and organoleptic value (vegan burger), developed through the substitution of animal proteins and lipids with plant-based constituents using innovative technologies, compared to a conventional burger, in apparently healthy subjects.

The study will be a randomized, cross-over, double blind clinical trial. The study sample will consist of 15 apparently healthy subjects aged 30-60 years, with a body mass index of ≥25 kg/m2 and a habitual red meat consumption of ≥3 times/week. Candidates will be excluded from the study on the basis of the following: i) presence of chronic diseases, such as diabetes mellitus, active cancer, cardiovascular, liver kidney, respiratory, gastrointestinal, chronic inflammatory and psychiatric diseases; ii) use of certain types of medication, i.e., immunosuppressants, anti-inflammatory drugs and cortisol, and dietary supplements, i.e., protein, amino acids, fatty acids, dietary fiber, probiotics and prebiotics (other prescribed medications and micronutrient supplements will be allowed, provided that their reception will remain stable throughout the trial); iii) habitual excessive consumption of alcohol (>210 g and >140 g of ethanol per week for men and women, respectively), iv) currently being on a restrictive diet (e.g., weight loss or vegetarian diet) or any significant recent change (within 6 months) in lifestyle habits, and v) pregnancy and breastfeeding for women.

Participants will be randomized to consume 2 servings per week of either a conventional burger or a vegan burger (serving size: 150 g of raw product corresponding to 120 g of cooked product) for 4 weeks, with a 2-week wash-out period between the two interventions. Randomization will be performed by a researcher with no clinical involvement in the study and will be blind to all members of the research team.

All burger products will be prepared by a certified food industry (Hellenic Catering S.A.) based on current food safety legislation and quality assurance specifications. The conventional burger will be the animal(beef)-based burger already produced and marketed by the company, while the experimental burger (vegan burger) will be developed using innovative technologies from plant-based products, such as proteins and dietary fibers from legumes and edible strains of basidiomycetes, lipids of plant origin rich in n-3 polyunsaturated fatty acids and other bioactive components. The development of the methodologies for the isolation of the raw materials will be performed by the Laboratory of Design and Process Analysis, School of Chemical Engineering, National Technical University of Athens and the Laboratory of Biotechnology, Department of Biological Applications & Technology, University of Ioannina. The development of the experimental vegan burger to be used in the dietary intervention will take place in a pilot unit of Hellenic Catering S.A. A product preparation will be designed with the incorporation of vegetable proteins from meat analogues, with the aim of the final product composition meeting the desired technical characteristics of structure and texture as well as the organoleptic characteristics of a burger. An appropriate mold and molding machine will be selected to shape the product, and appropriate packaging, preservation and processing methods (e.g., sock freezing, chilling, cooking) will be utilized. The two burger products will have a common shape and organoleptic characteristics (odor, texture and taste).

Participants will be given additional instructions to maintain their usual dietary intake, physical activity level, prescribed medications and dietary supplements, as well as to refrain from any weight loss effort throughout the study. The study physician will be on a weekly contact with each participant to systematically record potential side-effects and will be in charge of terminating the intervention if needed. Participants' adherence to the intervention will be assessed through weekly self-monitoring diaries, in which subjects will record the day of consumption, the quantity and the cooking method of the burger products, along with other dietary characteristics and the use of medications and dietary supplements. Participants will be evaluated at the start and at the end of each intervention period (total of 4 evaluations) in terms of anthropometric indices, body composition, and lifestyle habits (diet and physical activity) through validated questionnaires, while fasting blood and first-morning urine samples will be taken to determine laboratory parameters (glucose metabolism indices, lipidemic profile, liver enzymes, inflammatory and oxidative stress markers, etc.). All biological samples will be collected and analyzed in the Laboratory of Clinical Nutrition and the Laboratory of Biology, Biochemistry, Physiology and Microbiology, Department of Nutrition and Dietetics, Harokopio University of Athens, by experienced personnel.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-60 years old
2. Body mass index ≥25 kg/m2
3. Habitual red meat consumption ≥3 portions/week (1 portion: 120 g cooked meat)

Exclusion Criteria:

1. Presence of chronic diseases, such as diabetes mellitus, active cancer, cardiovascular, liver kidney, respiratory, gastrointestinal, chronic inflammatory and psychiatric diseases
2. Reception of immunosuppressant, anti-inflammatory or cortisol medication,
3. Intake of protein, amino acid, fatty acid, dietary fiber, probiotic and prebiotic supplements
4. Habitual excessive alcohol consumption, i.e., >210 g and >140 g of ethanol per week for men and women, respectively
5. Currently being on a restrictive diet (e.g., weight loss or vegetarian diet) or any significant recent change (within 6 months) in lifestyle habits
6. Pregnancy and breastfeeding for women

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in homeostasis model of assessment - insulin resistance (HOMA-IR) at 4 weeks | 0 (baseline) and 4 weeks
  HOMA-IR will be calculated based on fasting glucose and fasting insulin levels through the Mathews equation. Fasting glucose and insulin will be measured in serum via a photometric method in a biochemical analyzer.
Change from baseline in total cholesterol at 4 weeks | 0 (baseline) and 4 weeks
  Total cholesterol will be measured in serum via a photometric method in a biochemical analyzer.
Change from baseline in low-density lipoprotein (LDL) cholesterol at 4 weeks | 0 (baseline) and 4 weeks
  LDL cholesterol will be measured in serum via a photometric method in a biochemical analyzer.
Change from baseline in high-density lipoprotein (LDL) cholesterol at 4 weeks | 0 (baseline) and 4 weeks
  HDL cholesterol will be measured in serum via a photometric method in a biochemical analyzer.
Change from baseline in triglycerides at 4 weeks | 0 (baseline) and 4 weeks
  Triglycerides will be measured in serum via a photometric method in a biochemical analyzer.
Change from baseline in uric acid at 4 weeks | 0 (baseline) and 4 weeks
  Uric acid will be measured in serum via a photometric method in a biochemical analyzer.
Change from baseline in urea at 4 weeks | 0 (baseline) and 4 weeks
  Urea will be measured in serum via a photometric method in a biochemical analyzer.
Change from baseline in high sensitivity C-reactive protein (hsCRP) at 4 weeks | 0 (baseline) and 4 weeks
  hsCRP will be measured in serum via an enzyme-linked immunoassay.
Change from baseline in systolic blood pressure (SBP) at 4 weeks | 0 (baseline) and 4 weeks
  SBP will be measured with an automatic device operating on the oscillometric principle.
Change from baseline in diastolic blood pressure (DBP) at 4 weeks | 0 (baseline) and 4 weeks
  DBP will be measured with an automatic device operating on the oscillometric principle.

SECONDARY OUTCOMES:
Change from baseline in hematocrit at 4 weeks | 0 (baseline) and 4 weeks
  Hematocrit will be measured in a hematology analyzer.
Change from baseline in iron at 4 weeks | 0 (baseline) and 4 weeks
  Iron will be measured in serum via a photometric method in a biochemical analyzer.
Change from baseline in ferritin at 4 weeks | 0 (baseline) and 4 weeks
  Ferritin will be measured in serum via a chemiluminescent immunoassay in a biochemical analyzer.
Change from baseline in total iron binding capacity at 4 weeks | 0 (baseline) and 4 weeks
  Total iron binding capacity will be measured in serum via a photometric method in a biochemical analyzer.
Change from baseline in albumin at 4 weeks | 0 (baseline) and 4 weeks
  Albumin will be measured in serum via a photometric method in a biochemical analyzer.
Change from baseline in alanine aminotransferase (ALT) at 4 weeks | 0 (baseline) and 4 weeks
  ALT will be measured in serum via a photometric method in a biochemical analyzer.
Change from baseline in gamma-glutamyl transferase (GGT) at 4 weeks | 0 (baseline) and 4 weeks
  GGT will be measured in serum via a photometric method in a biochemical analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Tzortzis Nomikos, PhD, Principal Investigator — Department of Nutrition and Dietetics, School of Health Sciences and Education, Harokopio University; Smaragdi Antonopoulou, PhD, Study Chair — Department of Nutrition and Dietetics, School of Health Sciences and Education, Harokopio University; Elizabeth Fragopoulou, PhD, Study Chair — Department of Nutrition and Dietetics, School of Health Sciences and Education, Harokopio University; Meropi Kontogianni, PhD, Study Chair — Department of Nutrition and Dietetics, School of Health Sciences and Education, Harokopio University; Michael Georgoulis, PhD, Study Director — Department of Nutrition and Dietetics, School of Health Sciences and Education, Harokopio University
Locations (1):
- Department of Nutrition and Dietetics, School of Health Sciences and Education, Harokopio University, Kallithea, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be shared to investigators for the purpose of data meta-analysis, provided that the proposed use has been approved by the Study Principal Investigator. Proposals should be directed to tnomikos@hua.gr. To gain access, data requestors will need to sign a data access agreement.